CLINICAL TRIAL: NCT06735001
Title: Identification of the Metabolic Signature of Atrial Fibrillation for Personalized Prevention
Acronym: IMAGE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2024/01
Record Dates: First submitted 2024-11-21; First posted 2024-12-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; prevention; biomarkers; cardiac metabolism
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: prospective multicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with FA (Other): Patient with a documented Fibrillation Atrial within the last 18 months
  Interventions: Procedure: FA ablation; Biological: Lab test
- Patients without FA (Other): Patient without Fibrillation Atrial
  Interventions: Biological: Lab test

INTERVENTIONS:
Procedure: FA ablation — Ablation of the FA
  Arms: Patients with FA
Biological: Lab test — Blood collection

SUMMARY:
Atrial fibrillation (AF) is a major public health problem. The efficacy of the existing techniques is limited in the more aggressive forms. It is therefore necessary to develop approaches, in particular the identification of relevant biomarkers, to prevent the onset, recurrence or progression of AF in at-risk patients. The objective of this study is to describe the longitudinal metabolic and biomolecular signature of AF in patients eligible for cardiac ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major public health problem. Its prevalence exceeds 2%. The main aim of drug treatment is to prevent the onset of stroke and heart failure, but side effects often require discontinuation, and contraindications limit their use. Rhythm control strategies based on catheter ablation have led to significant progress in incident AF, improving quality of life. Nevertheless, the efficacy of these techniques is limited in the more aggressive forms. Significant recurrence rates are reported one year after ablation, and access to them is often reserved for symptomatic patients due to their invasive and costly nature.

It is therefore necessary to develop approaches to prevent the onset, recurrence or progression of AF in at-risk patients. While the pathophysiology of AF involves metabolic remodelling that can be observed in animal and human models, no clinically relevant metabolites have been identified as biomarkers of the risk of AF onset or progression, with a view to preventive and personalized management.

In response to this unmet need, this project aims to develop a method for assessing the risk of AF recurrence, combining the identification of a metabolic signature of the arrhythmia and the patient, with a machine learning approach to aggregate conventional risk factors and metabolic biomarkers. A longitudinal clinical study will be conducted on patients scheduled for AF ablation, to monitor changes in their metabolic signature over 12 months, in parallel with arrhythmia progression. Using machine learning, the study team will establish and validate a classifier retrospectively stratifying patients with or without recurrent AF, and compare this method with canonical risk stratification. This will enable to consider personalized management of patients at risk of recurrence, with the aim of reducing human and economic costs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, all genders, and ethnic origins
* Free, informed, and written consent signed
* Person affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Age < 18 years
* Lack of informed consent
* Gestating women (pregnancy test carried out as part of care for FA patients, contraception, or menopause for women in control groups)
* Persons under administrative or judicial protection
* Endocarditis or pericarditis in progress or within the 3 last months
* Active tumor pathology (benign or malignant)
* Chronic inflammation or autoimmune disease
* Chronic liver disease
* Myocardial infarction within the last 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Biomarkers T1 | Day 0
  The individuation of biomarkers uniquely present in AF patients - compared to control groups.
Biomarkers T2 | Day 1
  The individuation of biomarkers uniquely present in AF patients - compared to control groups.
Biomarkers 2 | 12 months
  The identification of biomarkers predictive of the risk of AF recurrence

SECONDARY OUTCOMES:
Algorithm | Month 12
  Identification of the machine learning algorithm with the best predictive performance for AF recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DERVAL, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: Undecided